CLINICAL TRIAL: NCT04555681
Title: Study of the Periodontal Microbiota in Gingival Cicatricial Pemphigoid Patients. Bicentric Pilot Study .
Brief Title: Study of the Periodontal Microbiota in Gingival Cicatricial Pemphigoid Patients. Bicentric Pilot Study.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20-PP-01; 2020-A01670-39 (Registry Identifier: ID RCB)
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Preservation of bacteriological samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Collection of subgingival dental plaque — Identification and quantification using q-PCR of the 21 bacteria most frequently found in the dental plaque (including the periopathogenic bacteria) and Candida albicans.

SUMMARY:
In patients with gingival cicatricial pemphigoid (CP), clinical experience has shown that periodontal treatment is beneficial in addition to medical treatment, because the latter does not always allow optimal gingival healing. However in practice, the basic periodontal treatment, combining subgingival scaling and debridement, may be insufficient especially for severe forms of erosive gingivitis. Therefore, a better knowledge of the periopathogenic flora in such patients would facilitate the implementation of a more appropriate and efficient periodontal therapy. In order to meet this objective, we propose a qualitative analysis of the periodontal microbiota in case of gingival CP via a bi-centric observational microbiological pilot study.

DETAILED DESCRIPTION:
In gingival cicatricial pemphigoid (PC) patients, clinical experience has shown that periodontal treatment is beneficial in addition to medical treatment, because the latter does not always allow optimal gingival healing. When the tissue remains erosive despite the systemic treatment, and/or local, anti-inflammatory and/or immunosuppressive, patients frequently report persistent oral discomfort that restricts their diet as well as difficulties in brushing their teeth. Accumulation of dental plaque, organized in bacterial biofilms, therefore becomes inavoidable. However, due to their increasing development, studies have revealed that this dysbiotic periodontal microbiota promotes the growth of virulent, anaerobic, proteolytic bacteria, with high invasive and deleterious properties for periodontal tissues. Furthermore, this process would be amplified in the presence of gingival erosive zones. By eliminating the infectious periodontal gateway, periodontal therapy should allow : i/to restore oral comfort ii/ to prevent any systemic oral infectious complications that may affect the general condition of patients or counteract the effects of drug therapies iii/ to limit the aggravation of concomitant periodontal diseases, and therefore the risk of tooth loss. However in practice, the basic periodontal treatment, combining subgingival scaling and debridement does not systematically meet these objectives. One explanation may be found in the quality of dental bacterial biofilms not yet determined for autoimmune bullous diseases. The main objective of our descriptive observational pilot study, was therefore to study the composition of the periopathogenic flora in patients with gingival CP in order to facilitate the implementation of a more appropriate and efficient periodontal therapy. The secondary objectives were to establish a potential correlation between the composition of this flora and the quality of oral life, the severity of the erosive gingival damage, whether or not to initiate medical treatment, and whether or not there is an underlying periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old) consultant in the odontology department of Saint Roch Hospital in Nice or Henri Mondor in Créteil, with erosive gum expression PCs, in acute or stabilization phase after the introduction of medical treatment, regardless of their general health conditions but without eye damage and laryngée. The diagnosis of PC must have been certified by a hospital dermatologist
* Patients affiliated with Social Security.
* Informed consent signed.

Exclusion Criteria:

* Antibiotic therapy and antifungal 3 months before the study.
* Mechanical periodontal treatment 3 months before the study.
* Refusal of the patient to participate in the study.
* People under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (over 18 years old) consultant in the odontology department of Saint Roch Hospital in Nice or Henri Mondor in Créteil, with erosive gum expression PCs
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Identification and quantification of candida albicans in subgingival dental plaque | The day of patient inclusion.
  The day of patient inclusion. Collection of subgingival dental plaque. Identification and quantification using q-PCR of Candida albicans.
Identification and quantification of 21 bacteria in subgingival dental plaque | The day of patient inclusion.
  Identification and quantification using q-PCR of the 21 bacteria most frequently The day of patient inclusion. Collection of subgingival dental plaque.
  Identification and quantification using q-PCR of the 21 bacteria most frequently found in the dental plaque (including the periopathogenic bacteria)

SECONDARY OUTCOMES:
Assessement of pain | The day of patient inclusion.
  Assessment of the intensity of oral pain using an analog visual scale (AVS).
Assessment of oral quality | The day of patient inclusion.
  Assessment of oral quality of life using the OHIP-14 score (Oral Health Impact Profile 2014). Periodontal clinical status : dental formula, assessment of tooth mobility, plaque index, gingival inflammation index, periodontal pocket probing, measurement of recessions, extent of erosive gingivitis.
Quantify alveolysis and severity. | The day of patient inclusion.
  Standard X-ray assessment (panoramic X-ray) to determine whether or not alveolysis is present and quantify its severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Myriem DRIDI, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CHU de Nice, Nice, CHU de NICE
  - HEnry Mondor, Paris

IPD SHARING:
Plan to Share IPD: No